CLINICAL TRIAL: NCT03483350
Title: Comparison of Granisetron Versus Midazolam and Thier Combination for Prophylaxis of Postoperative Nausea and Vomiting in Laparoscopic Surgery in Children
Brief Title: Comp Granisetron Midazolam Comb in Lap Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wesam Nashat Ali, Lecturer of anesthesiology Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Gmpl
Record Dates: First submitted 2018-02-13; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Granisetron; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1- 1st group (Experimental): 1- 1st group will include 30 patients will receive intravenous granisetron 10 μg/kg after induction of anesthesia and before start of surgery
  Interventions: Drug: Granisetron
- 2- 2nd (Experimental): 2- 2nd group will include 30 patients will receive intravenous midazolam 50 μg/kg after induction of anesthesia and before start of surgery
  Interventions: Drug: Midazolam
- 3- 3rd group (Experimental): 3- 3rd group will include 30 patients will receive combination intravenous granisetron 5 μg/kg with midazolam 25 μg/kg after induction of anesthesia and before start of surgery
  Interventions: Drug: Granisetron; Drug: Midazolam

INTERVENTIONS:
Drug: Granisetron — Ampoule
  Arms: 1- 1st group; 3- 3rd group
Drug: Midazolam — Ampoule
  Arms: 2- 2nd; 3- 3rd group

SUMMARY:
Postoperative nausea and vomiting (PONV) is one of the most common complications of general anesthesia in pediatrics. Pediatric rates of nausea and vomiting are approximately double those of adult patients.

The physiology of PONV is complex and not perfectly understood. According to our current model, the brain structures involved in the pathophysiology of vomiting are distributed throughout the medulla oblongata of the brainstem, not centralized in an anatomically defined 'vomiting centre. Such structures include the chemoreceptor trigger zone (CRTZ), located at the caudal end of the fourth ventricle in the area postrema, and the nucleus tractus solitarius (NTS), located in the area postrema and lower pons.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is one of the most common complications of general anesthesia in pediatrics. Pediatric rates of nausea and vomiting are approximately double those of adult patients.

The physiology of PONV is complex and not perfectly understood. According to our current model, the brain structures involved in the pathophysiology of vomiting are distributed throughout the medulla oblongata of the brainstem, not centralized in an anatomically defined 'vomiting centre. Such structures include the chemoreceptor trigger zone (CRTZ), located at the caudal end of the fourth ventricle in the area postrema, and the nucleus tractus solitarius (NTS), located in the area postrema and lower pons. The CRTZ receives input from vagal afferents in the gastrointestinal tract, and it can also detect emetogenic toxins, metabolites, and drugs circulating in the blood and cerebrospinal fluid due to its lack of the bloodbrain barrier. Multiple neurotransmitter pathways are implicated in the physiology of nausea and vomiting. Enterochromaffin cells in the gastrointestinal tract release serotonin, and the vagus nerve communicates with the CRTZ via 5-HT3 receptors. The CRTZ communicates with the NTS primarily via dopamine-2 (D2) receptors.

PONV may increase hospital expenditure by prolongation of hospital stay, and management of vomiting related complications such as dehydration, electrolyte disturbances, and pulmonary aspiration. Pediatric laparoscopic surgery is commonly associated with higher incidence of PONV. Mixtures of different classes of antiemetics have been used successfully to decrease the incidence of PONV but there was no agreement on the optimal combination. Granisetron a newer 5-HT3 antagonist has stronger receptor binding and has been found to be more potent and longer acting as antiemetic for preventing postoperative nausea and vomiting following laparoscopic surgery. Midazolam is commonly used as a premedication to relief anxiety. Midazolam given intravenously before the end of surgery was effective in decreasing the incidence of PONV. sub-hypnotic dose of midazolam was suggested that have a role in the management of PONV.

ELIGIBILITY:
Inclusion Criteria:

* This study will include children, scheduled for elective Laparoscopic surgery
* Age 4-12 years
* ASA I or II

Exclusion Criteria: Patients will be excluded who meet these criteria

* Patient refusal
* Any contraindication of laparoscopic surgery;as personal history of seizures, peripheral neurologic diseases, cardiac arrhythmias, liver disease, renal dysfunction and cardiac conduction abnormalises
* Known allergy to the drugs included in the study

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Vomiting score | for48hours(two day)
  Have you vomited?
  0 - No, 1 - Once, 2 - Twice, 3 - Three or more time

SECONDARY OUTCOMES:
Nausea score | for48hours(two day)
  Have you experienced feeling of nausea (an unsettled feeling in the stomach and slight urge to vomit)
  0-No 1-Yes

REFERENCES:
- [Background] Gan TJ, Meyer T, Apfel CC, Chung F, Davis PJ, Eubanks S, Kovac A, Philip BK, Sessler DI, Temo J, Tramer MR, Watcha M; Department of Anesthesiology, Duke University Medical Center. Consensus guidelines for managing postoperative nausea and vomiting. Anesth Analg. 2003 Jul;97(1):62-71, table of contents. doi: 10.1213/01.ane.0000068580.00245.95. PMID 12818945